CLINICAL TRIAL: NCT05491889
Title: Outcome of Hepatocellular Carcinoma Patients With Portal Vein Thrombosis After Trans-Arterial Chemo Embolization
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alshaimaa Eid, Resident doctor, Assiut University
Other Study IDs: 17101837
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HCC patients with PPVT after TACE: determine frequency of short-term mortality (< 3month) among HCC patients with PPVT after TACE, and to explore its predictors.
  Interventions: Biological: trans arterial chemoembolization

INTERVENTIONS:
Biological: trans arterial chemoembolization — trans arterial chemoembolization in patient with partial portal vein thrombosis

SUMMARY:
Hepatocellular carcinoma (HCC) is the fifth most common neoplasm worldwide and the third most frequent cause of death from cancer in the world. Hepatocellular carcinoma is responsible for significant morbidity and mortality in cirrhosis. Most cases of HCC occur in the setting of cirrhosis and, therefore, prognosis is determined not only by factors related to the tumor but also by factors related to cirrhosis (1).

According to previous reports, the incidence of HCC with partial portal vein thrombosis (PVTT) ranges between 44% and 62.2%. HCC associated with PVTT has a poor prognosis. It may lead to intrahepatic metastasis, liver dysfunction, and portal hypertension. The median overall survival for HCC patients with untreated PVTT is only 2.7 months (2).

It was suggested that HCC with PVTT should be classified as stage C based on Barcelona Clinic Liver Cancer; it is no longer surgically treatable. Compared with conservative treatment, TACE is a safe and effective therapy for such cases. However, this modality for treatment might be associated with mortality (3).

As far as we know, there is no studies of short-term survival in patients with HCC and PVT after TACE in our locality.

Our study aims to determine frequency of short-term mortality (< 3month) among HCC patients with PPVT after TACE, and to explore its predictors.

DETAILED DESCRIPTION:
Type of the study:cohort study Study Setting: Assiut University Hospitals

Sample Size Calculation:

Total coverage sample technique will be applied in the current study where all patients who are fulfilling inclusion criteria during the study period will be included.

Study tools (in detail, e.g., lab methods, instruments, steps, chemicals, …):

For all the study patients, clinical evaluation (including demographic data and body mas index), laboratory investigations (including liver and kidney chemistry, INR, and complete blood picture), and imaging studies (including abdominal ultrasonography, doppler ultrasonography, and contrast computed tomography) will be provided.

CTP and MELD scores will be calculated.

Data management and analysis (Details needed):

Data collection: will include patients between 2015 and 2023. Computer software

Statistical tests:

Based on short term survival, eligible patients will be subdivided into two groups either survivors or non-survivors. Continuous data will be given in form of mean (SD) and compared by Student t test while nominal data will be expressed as frequency (percentage) and chi square test is used for such data.

Overall survival analysis will be done by Kaplan Meier survival curve. Logistic regression analysis will be applied to determine the possible predictors for short term mortality.

Level of confidence is kept at 95% and hence, p value is considered significant if < 0.05. Analysis of data will be done by SPSS 28 software

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* HCC was diagnosed based on contrast imaging
* PPVT was diagnosed based on abdominal Duplex

Exclusion Criteria:

* Age < 18 years old
* Complete PVT
* Any previous therapy for HCC
* Extrahepatic concomitant malignancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patient with hepatocellular carcinoma with partial portal vein thrombosis
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
mortality | 3 months
  frequency of short term mortality

IPD SHARING:
Plan to Share IPD: No
all researcher will be blinded about data collection from other researchers.

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Zhang ZM, Lai EC, Zhang C, Yu HW, Liu Z, Wan BJ, Liu LM, Tian ZH, Deng H, Sun QH, Chen XP. The strategies for treating primary hepatocellular carcinoma with portal vein tumor thrombus. Int J Surg. 2015 Aug;20:8-16. doi: 10.1016/j.ijsu.2015.05.009. Epub 2015 May 27. PMID 26026424
- [Background] Xiang X, Lau WY, Wu ZY, Zhao C, Ma YL, Xiang BD, Zhu JY, Zhong JH, Li LQ. Transarterial chemoembolization versus best supportive care for patients with hepatocellular carcinoma with portal vein tumor thrombus：a multicenter study. Eur J Surg Oncol. 2019 Aug;45(8):1460-1467. doi: 10.1016/j.ejso.2019.03.042. Epub 2019 Apr 12. PMID 31005471